CLINICAL TRIAL: NCT03630627
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Rising Dose Study to Explore the Safety, Tolerability, and Pharmacokinetics of Intravenous Doses of SB26 in Healthy Volunteers
Brief Title: A Phase I Study of SB26 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB26-1001
Record Dates: First submitted 2018-04-05; First posted 2018-08-15 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SB26 for Part 1 (Experimental): SB26: various single doses, administered to various cohorts
  Interventions: Drug: SB26
- SB26 for Part 2 (Experimental): SB26: various multiple doses, administered to various cohorts
  Interventions: Drug: SB26
- Placebo for Part 1 (Placebo Comparator): SB26 matching placebo: various single doses, administered to various cohorts
  Interventions: Drug: Placebo
- Placebo for Part 2 (Placebo Comparator): SB26 matching placebo: various multiple doses, administered to various cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB26 — SB26 administered intravenously
  Other Names: TAK-671
  Arms: SB26 for Part 1; SB26 for Part 2
Drug: Placebo — Placebo administered intravenously
  Other Names: SB26/TAK-671 matching placebo
  Arms: Placebo for Part 1; Placebo for Part 2

SUMMARY:
This study is a Phase I, randomized double-blind, placebo-controlled (within a dose group), single and multiple rising dose study of the intravenous administration of SB26 in healthy volunteers.

DETAILED DESCRIPTION:
The study includes two Parts; Part 1 includes the FiH exposure and SRD and Part 2 is the MRD. Approximately 58 subjects will be enrolled in the study. New subjects will be recruited for each cohort in both Parts. The SRD Part will include 5 or more dose levels and the MRD Part will include 3 or more dose levels; additional dose level(s) may be added based on emerging safety and PK data from prior cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the Investigator, the subject is capable of understanding and complying with protocol requirements.
2. The subject signs and dates a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures.
3. The subject is willing to comply with study procedures and restrictions.
4. The subject is a healthy adult man or woman of non-childbearing potential.
5. The subject is aged 18 to 65 years, inclusive, at the time of informed consent.
6. The subject weighs at least 50 kg and has a body mass index from 18 to 32 kg/m2, inclusive, at Screening.
7. If the subject is a male who is non-sterilized and who is sexually active with a female partner of childbearing potential, agrees to use adequate contraception from signing of ICF throughout the duration of the study until 60 days (i.e., estimated > 5 half-lives) after the last dose of study drug(s).
8. The subject is a non-smoker or ex-smoker who has not used tobacco- or nicotine-containing products (e.g., nicotine patch) for at least 6 months prior to first administration of study drug (Day 1) and who has had a negative urine cotinine at Screening and Check-in (Day -1).

Exclusion Criteria:

1. The subject has received any investigational compound or medication within 30 days or five half-lives, whichever is the longest, prior to the first intended dose of study drug.
2. The subject is a study site employee, immediate family member thereof, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, or sibling) or may consent under duress.
3. The subject has a known hypersensitivity to any component of the formulation of SB26, or has had clinically significant infusion-related reactions to any prior biologic drug unless it can be established that the reaction was due to components not present in the formulation of SB26.
4. The subject has a positive urine result for drugs of abuse at Screening or Check-in (Day -1).
5. The subject has a history of drug abuse or a history of alcohol abuse (defined as drinking alcoholic beverages of more than 21 units per week for males and 14 units per week for females; 1 unit = 14 g of pure alcohol, e.g., 1 unit = 250 mL of beer, 25 mL of spirits or one glass [125 mL] of wine) within 1 year prior to Screening.
6. If male, the subject intends to father a child or to donate sperm during the course of this study until 60 days after the last dose of study drug.
7. The subject has evidence of current or recent (within 6 months prior to Screening) disease that, in the opinion of the Investigator, may pose additional risks to the subject or confound the assessment of safety and tolerability. This should be discussed with the Sponsor's medical representative if there is uncertainty about the suitability of the subject.
8. The subject has a history of cancer, except basal cell carcinoma or cervical carcinoma in situ that has been treated and in remission for at least 5 years prior to Screening.
9. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus at Screening.
10. The subject has poor peripheral venous access at Screening or Check in (Day -1).
11. The subject has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis) in the 30 days prior to Screening.
12. The subject has an electrocardiogram (ECG) showing a clinically significant abnormality at Screening or Check-in (Day -1). Entry of any subject with an abnormal but not clinically significant ECG must be approved, and documented by signature of the Principal Investigator or a medically qualified sub-Investigator.
13. The subject's ECG has a QT interval with Fridericia correction method > 450 msec for male, > 470 msec for female or a PR interval outside the range 120 to 220 msec, confirmed on repeat testing within a maximum of 30 minutes, at Screening or Check-in (Day -1).
14. The subject has a sustained resting heart rate outside the range 40 to 100 beats per minute, confirmed on repeat testing within a maximum of 30 minutes, at Screening or Check-in (Day -1).
15. The subject has systolic blood pressure > 140 or < 90 mmHg or a diastolic blood pressure > 90 or < 50 mmHg at Screening or Check-in (Day -1). One repeat testing is allowed at Screening and Check-in (Day -1)
16. The subject has any other abnormal laboratory values at Screening or Check-in (Day -1), confirmed upon repeat testing, that suggest a clinically significant underlying disease per the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAE | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Experience at least 1 treatment-emergent adverse event
Incidence of AE leading to discontinuation | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Discontinue due to adverse event
Abnormal hematology parameters | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal hematology parameters. The following parameters will be analyzed: White blood cell, red blood cell, hemoglobin, platelet count.
Abnormal serum chemistry parameters | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal serum chemistry parameters. The following parameters will be analyzed: Blood urea nitrogen, creatinine, total protein, albumin, alanine transaminase, aspartate transaminase.
Abnormal coagulation parameters | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal coagulation parameters. The following parameters will be analyzed: Prothrombin time, activated partial thromboplastin time.
Abnormal urinalysis parameters | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal urinalysis parameters. The following parameters will be analyzed: Protein, glucose, urobilinogen, bilirubin.
Abnormal blood pressure | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal blood pressure. Systolic blood pressure (SBP), diastolic blood pressure (DBP) will be measured in a supine position after at least 5 minutes of rest.
Abnormal heart rate | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal heart rate. It will be measured in a supine position after at least 5 minutes of rest.
Abnormal body temperature | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal body temperature. It will be measured in a supine position after at least 5 minutes of rest.
Abnormal ECG | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Meet the criteria for markedly abnormal 12-lead ECG parameter. QT interaval with Fridericia correction method (QTcF) value will be measured in a supine position after at least 10 minutes of rest.

SECONDARY OUTCOMES:
Cmax | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Maximum observed serum concentration
tmax | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Time to reach Cmax
AUClast | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Area under the curve from the time of dosing to the time of the last measurable concentration
Vd | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Volume of distribution
CL | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Total body clearance
t1/2 | Part 1: From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Terminal half-life
AUCinf | Part 1: From Day 1 until Day 50
  Area under the curve from the time of dosing extrapolated to infinity
Accumulation index | Part 1: From Day 1 until Day 50
  Predicted using terminal rate constant and dosing interval
AUCtau | Part 2: From Day 1 until Day 71
  Area under the serum concentration-time curve over the dosing interval
Accumulation ratio | Part 2: From Day 1 until Day 71
  Calculated using systemic exposure at first dosing and last dosing
Cmin | Part 2: From Day 1 until Day 71
  Minimum observed concentration
Incidence of ADA | From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Incidence of anti-drug antibody
Titer of ADAs | From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Titer of anti-drug antibodies to SB26
Incidence of NAb | From Day 1 until Day 50; Part 2: From Day 1 until Day 71
  Incidence of neutralizing antibody to SB26

CONTACTS AND LOCATIONS:
Overall Officials: David Han, M.D., Principal Investigator — California Clinical Trials Medical Group, a division of PAREXEL International
Locations (1):
- PAREXEL International, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No